CLINICAL TRIAL: NCT00726817
Title: The Effects of Butyrate Enemas on Visceral Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Robert-Jan Brummer, Prof, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MEC 06-3-020
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2008-07

CONDITIONS: Visceral (Hyper)Sensitivity
Keywords: butyrate, visceral perception, compliance
MeSH Terms: conditions — Patient Compliance | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): enemas, once daily, containing saline
  Interventions: Drug: Butyrate
- 2 (Experimental): enemas, once daily, containing 50mM butyrate
  Interventions: Drug: Butyrate
- 3 (Experimental): enemas, once daily, containing 100mM butyrate
  Interventions: Drug: Butyrate

INTERVENTIONS:
Drug: Butyrate

SUMMARY:
During this double blind, placebo controlled, randomised cross over study, healthy volunteers received an enema once daily for one week containing either placebo (saline), 50mM butyrate or 100mM of butyrate. Before and directly after each test period a barostat protocol was performed to measure parameters for visceral perception.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* age, under 18 or over 65
* use of pre- or probiotics during study and 3 months previous to study
* previous bowel complaints
* gastrointestinal disease or abdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert-Jan Brummer, Prof, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands